CLINICAL TRIAL: NCT03520777
Title: A Pilot Study of Creative Arts Interventions for Neurology Inpatients in the Epilepsy Monitoring Unit and the Headache Service
Brief Title: A Pilot Study of Creative Arts Interventions for Neurology Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Lara K. Ronan, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 30498
Record Dates: First submitted 2018-04-13; First posted 2018-05-11 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Epilepsy; Migraine
MeSH Terms: conditions — Epilepsy; Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artist Intervention (Other): One of the three artists (visual artist, music therapist, creative writer) will work with subjects for up to 90 minutes.
  Interventions: Other: Art Intervention

INTERVENTIONS:
Other: Art Intervention — Type of artist intervention will be determined by the subject and the assigned artist.

SUMMARY:
The purpose of the study is to assess the feasibility of a Creative Artists Program intervention with epilepsy and headache patients admitted to Dartmouth-Hitchcock Medical Center for care by the Department of Neurology.

DETAILED DESCRIPTION:
Qualifying patients admitted to Epilepsy monitoring or Headache treatment will be approached for participation in the study. Patients who consent to the study will be given a chance to work with one of three creative artists (visual artist, creative writer, therapeutic musician). The artist will be selected according to a pre-determined schedule, and the arts intervention may last up to 90 minutes. Subjects will be asked to complete study questionnaires before and after the arts intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 18 years
2. Diagnosis of refractory chronic epilepsy, status migrainosus, or chronic daily headache
3. Elective admission to the Dartmouth-Hitchcock Medical Center Epilepsy monitoring unit or Headache service
4. Capable of giving informed consent

Exclusion Criteria:

1. Active psychiatric illness that prohibits safe visitation by artists
2. Impairment of vision or hearing that would prohibit able to participate with participation in instructions necessary for the interventions.
3. Active general medical condition that would impair consciousness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting a creative arts intervention study | Through study completion, approximately 1 year
  The feasibility of the creative intervention will be determined by the completion rates of the initial intervention attempts. If less than 50% of patients complete the intervention it will be deemed unfeasible in the current format.

SECONDARY OUTCOMES:
Change in patient anxiety before and after the intervention | Each patient will be assessed at baseline (Day 1) and after the intervention (approximately Day 3 - 21).
  Change in anxiety level will be calculated, based on patient questionnaire responses, following the creative intervention.
Change in patient distress before and after the intervention | Each patient will be assessed at baseline (Day 1) and after the intervention (approximately Day 3 - 21).
  Change in distress level will be calculated, based on patient questionnaire responses, following the creative intervention.
Change in patient depression before and after the intervention | Each patient will be assessed at baseline (Day 1) and after the intervention (approximately Day 3 - 21).
  Change in depression level will be calculated, based on patient questionnaire responses, following the creative intervention.
Change in frequency of as-needed pain medication use | Each patient as-needed medication use will be assessed after the arts intervention and until discharge from the hospital (approximately Day 3 - 21).
  As-needed pain medication utilization will be evaluated following the creative arts intervention through subject discharge.
Length of hospital stay | Each patient's admission duration (approximately 3 - 21 Days).
  Length of hospital stay will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States